CLINICAL TRIAL: NCT04020731
Title: Physiological Changes Exploration During the Hypnotic State (HYPNOTE)
Brief Title: Physiological Changes Exploration During the Hypnotic State
Acronym: HYPNOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC19.060
Record Dates: First submitted 2019-06-21; First posted 2019-07-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers
Keywords: Hypnosis; MEG; Auditory Evoked Magnetic Fields; Oscillatory activity; Networks
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Right-handed healthy volunteers (Experimental): Magnetoencephalography (MEG) records
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — several blocks of hypnosis including entry into a hypnotic state (= induction), the hypnotic trance and the exit from hypnosis (= reassociation).

SUMMARY:
Use of hypnosis for therapeutic purposes tends to spread. However, the neural mechanisms underlying hypnosis is still debated and no specific change has yet been associated with this state. In this context, it seems necessary to clarify its mechanisms and effects. Since hypnosis induces a change of consciousness state, the investigators hypothesize that this modification is accompanied by neural activity changes recordable with magnetoencephalography (MEG). The primary objective of this study is to identify neural activity changes during hypnotic trance in healthy volunteers.

DETAILED DESCRIPTION:
Since the 19th century, the potential changes induced by hypnosis have been investigated. Indeed, hypnosis induces a change on the usual state of conscious awareness. This state is accompanied by physiological changes, as cardiac and cerebral. However, although literature on the neural mechanisms underlying hypnosis increases, no specific activity change has been identified. Only the subjective judgment of hypnotherapist can assume the volunteer state. Considering that the use of hypnosis enhanced in the field of medical care, it is necessary to clarify and define it. This requires a better understanding of its mechanisms through the study of brain, heart and respiratory activities.

The aim of this clinical trial is to assess modifications of physiological signals (cardiac, respiratory and cerebral) before and during a session of hypnosis, to identify some biomarkers of the hypnotic trance. Therefore the cardiac, respiratory and cerebral activities will be recorded during hypnosis sessions and control state to compare the signals.

The MEG will be used to record brain activity due to its sensitivity in the very low and high frequencies, its temporal resolution and its robustness for the localization of neural origins. In accordance with the literature and preliminary results, changes in theta oscillations (4-8 Hz) will be assessed. In fact, these oscillations seem to be increased during the hypnotic state. So, it seems interesting to correlate these oscillations with potential changes in heart and/or respiratory rhythms.

This clinical trial is an open mono-centric study, performed on a cohort of healthy volunteers in which each subject is his own control (intra-subject control). The physiological parameters will be recorded and analyzed during three control states ("subject alone", "subject and hypnotherapist without communication" and "reading a book by the hypnotherapist"), and several blocks of hypnosis interleaved with an attentional task (stroop). All the collected parameters in these different conditions will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Right-handed
* Non-smoking
* Major participants
* Speaking fluent French
* No experience of hypnosis or other forms of meditation and relaxation
* Registered in the French social security scheme
* Signed informed consent

Exclusion Criteria:

* Contraindication to Magnetoencephalography (MEG) and/or Magnetic resonance imaging (MRI) : implanted material, claustrophobia,…
* Treatment that may impact physiological measures (psychotropic, cardiovascular,…)
* All categories of protected persons (Pregnant or lactating women, persons subject to a legal protection measure, persons deprived of their liberty by judicial or administrative decision)
* Smokers
* Persons with personality disorders or addictions / narcotic use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Neural activity changes recorded by magnetoencephalography (MEG) during hypnotic trance, in healthy volunteers. | 2 hours
  Oscillatory activity will be recorded by magnetoencephalography (MEG) : power averages of oscillations (delta, theta, alpha, beta and gamma) and phase values recorded during hypnotic trance will be compared to control conditions.

SECONDARY OUTCOMES:
Neural networks activity changes recorded by magnetoencephalography (MEG) during hypnotic trance, in healthy volunteers. | 2 hours
  Power average (Grad : fT²/Hz MAG : fT²/cm².Hz) of neuronal sources and correlations of sources activity for the Default Model Network (DMN) will be compared between hypnosis trance and control conditions.
Changes in auditory evoked magnetic fields (MAEF), recorded by magnetoencephalography (MEG) during hypnotic trance, in healthy volunteers. | 2 hours
  Global averages of MAEF (Grad : fT/(cm.√Hz) MAG : fT/√Hz) will be compared between hypnosis trance and control conditions.
Cardiac and respiratory changes in link to neural activity changes observed during the hypnotic trance | 2 hours
  Variations in heart rate and respiratory parameters (Hz) with neural activity changes previously described (ie: oscillatory activity, network activities (Grad : fT²/Hz MAG : fT²/cm².Hz) and MAEF (Grad : fT/(cm.√Hz) MAG : fT/√Hz)), will be compared between hypnosis trance and control conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Clinatec Cea/Chuga, Grenoble, France

REFERENCES:
- [Background] De Pascalis V, Ray WJ, Tranquillo I, D'Amico D. EEG activity and heart rate during recall of emotional events in hypnosis: relationships with hypnotizability and suggestibility. Int J Psychophysiol. 1998 Aug;29(3):255-75. doi: 10.1016/s0167-8760(98)00009-9. PMID 9666380
- [Background] Vanhaudenhuyse A, Laureys S, Faymonville ME. Neurophysiology of hypnosis. Neurophysiol Clin. 2014 Oct;44(4):343-53. doi: 10.1016/j.neucli.2013.09.006. Epub 2013 Oct 29. PMID 25306075
- [Background] Jensen MP, Adachi T, Hakimian S. Brain Oscillations, Hypnosis, and Hypnotizability. Am J Clin Hypn. 2015 Jan;57(3):230-53. doi: 10.1080/00029157.2015.985573. PMID 25928684
- [Background] Zeev-Wolf M, Dor-Ziderman Y, Goldstein A, Bonne O, Abramowitz EG. Oscillatory brain mechanisms of the hypnotically-induced out-of-body experience. Cortex. 2017 Nov;96:19-30. doi: 10.1016/j.cortex.2017.08.025. Epub 2017 Aug 31. PMID 28961523